CLINICAL TRIAL: NCT07390981
Title: Clinical Efficacy of Intradermal Acupuncture as an Adjunct to SSRI Dose Reduction or Discontinuation in Patients With Major Depressive Disorder and Its Mechanisms of Autonomic Nervous System Regulation
Brief Title: Intradermal Acupuncture for Assisting SSRI Dose Reduction in Major Depressive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Mingqi Tu, Doctor of Philosophy, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025KY394-1
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
Keywords: Intradermal Acupuncture; SSRIs; Heart Rate Variability
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SSRI Tapering Group (Active Comparator): Participants receive standard SSRI dose reduction or discontinuation under psychiatric supervision for 8 weeks.
  Interventions: Drug: Selective Serotonin Reuptake Inhibitors (SSRIs)
- SSRI Tapering + Sham Intradermal Acupuncture (Sham Comparator): Participants receive standard SSRI tapering combined with sham intradermal acupuncture for 8 weeks.
  Interventions: Drug: Selective Serotonin Reuptake Inhibitors (SSRIs); Procedure: Sham Intradermal Acupuncture
- SSRI Tapering + Intradermal Acupuncture (Experimental): Participants receive standard SSRI tapering combined with intradermal acupuncture for 8 weeks.
  Interventions: Drug: Selective Serotonin Reuptake Inhibitors (SSRIs); Procedure: Intradermal Acupuncture

INTERVENTIONS:
Drug: Selective Serotonin Reuptake Inhibitors (SSRIs) — Participants will receive only standard oral SSRI antidepressant dose reduction, with dosage adjustments determined by a specialist physician, for a duration of 8 weeks.
Procedure: Sham Intradermal Acupuncture — The sham intradermal needles are identical to the intradermal acupuncture needles in size, color, and material, with the needle body replaced by a thin silicone pad. The sham needles are applied to the selected acupoints and retained for 72 hours, followed by a 1-day rest period after removal. Acupoints: Shenmen (HT 7), Neiguan (PC 6), Sanyinjiao (SP 6), and Taichong (LR 3).
  Arms: SSRI Tapering + Sham Intradermal Acupuncture
Procedure: Intradermal Acupuncture — According to the location of the acupoints, intradermal acupuncture needles (φ0.20 × 1.5 mm or φ0.20 × 1.2 mm) are inserted vertically into the skin while avoiding blood vessels and retained for 72 hours, followed by a 1-day rest period after removal. During the retention period, participants are instructed to press the needles 3-4 times daily, with each stimulation lasting approximately 1 minute and an interval of 4 hours between sessions; the stimulation intensity is limited to the maximum level tolerated by the participant. Acupoints: Shenmen (HT 7), Neiguan (PC 6), Sanyinjiao (SP 6), and Taichong (LR 3).
  Arms: SSRI Tapering + Intradermal Acupuncture

SUMMARY:
This randomized controlled trial aims to evaluate the clinical efficacy of intradermal acupuncture as an adjunctive intervention to assist selective serotonin reuptake inhibitor (SSRI) dose reduction or discontinuation in adult patients with major depressive disorder (MDD). Participants receiving SSRIs and planning gradual dose reduction or discontinuation will be randomly assigned to one of three groups: SSRI tapering alone, sham intradermal acupuncture plus SSRI tapering, or intradermal acupuncture plus SSRI tapering. Clinical outcomes and autonomic nervous system function will be assessed to determine the effectiveness and potential mechanisms of intradermal acupuncture in facilitating SSRI reduction and alleviating withdrawal-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years

Diagnosis of major depressive disorder according to DSM-5

Currently receiving SSRI treatment and planning gradual dose reduction or discontinuation

Clear consciousness and ability to communicate normally

Willingness to participate and provide written informed consent

Exclusion Criteria:

* Severe uncontrolled primary medical conditions

Depression secondary to substances, medical illness, other psychiatric disorders (e.g., bipolar disorder, schizophrenia), or major bereavement

Active suicidal ideation

Pregnancy or lactation

Cognitive impairment

Bleeding disorders or allergy to adhesive materials

Participation in another clinical trial within the past month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
SSRI Dose Reduction Rate | Week 4, Week 8 (end of treatment), Week 12 (follow-up)
  Percentage reduction in SSRI dosage from baseline to each assessment point, calculated as:
  (Baseline dose - Post-treatment dose) / Baseline dose × 100%

SECONDARY OUTCOMES:
Change in SSRI Dosage | Week 4, Week 8, Week 12
  Absolute change in SSRI dose from baseline.
Depression Severity (HAMD-17) | Baseline, Week 4, Week 8, Week 12
  Clinician-rated Hamilton Depression Rating Scale (17-item).
Depression Severity (SDS) | Baseline, Week 4, Week 8, Week 12
  Self-Rating Depression Scale.
Antidepressant-Related Adverse Effects (SERS) | Baseline, Week 4, Week 8, Week 12
  Simpson Extrapyramidal Rating Scale.
Autonomic Nervous System Function (HRV Parameters) | Baseline, Week 8
  Time-domain and frequency-domain HRV parameters measured using 24-hour Holter monitoring.

IPD SHARING:
Plan to Share IPD: No